CLINICAL TRIAL: NCT06733714
Title: Association of Transcranial Alternating Current Stimulation with Digital Cognitive Training for Cognitive Remediation in Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Alzheimer's Association (Other); Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Rogerio Panizzutti, MD, PhD, Professor, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 38114820.3.0000.5263
Record Dates: First submitted 2024-12-05; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Cognitive Dysfunction; Alzheimer Disease; Mild Cognitive Impairment; Cognitive Decline; Frontotemporal Degeneration; Dementia; Dementia, Vascular; Lewy Body Disease; Beta-Amyloid; GFAP; Tau Protein
Keywords: tacs; nibs; transcranial alternate current stimulation; mild cognitive impairment; MCI; ALzheimer; Cognition; Elderly; Older Adults; Cognitive enhancement
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Dementia; Dementia, Vascular; Lewy Body Disease; Plaque, Amyloid; Frontotemporal Dementia; Spondylocostal Dysostosis 4, Autosomal Dominant | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: A random 5 digits password will be given to the care provider. This password will make the stimulation device enter SHAM mode or true stimulation mode, without the care provider or the patient knowing which mode it will be in.
  The SHAM mode has the Ramp up and Ramp down periods, so the participant allocated in the control-SHAM group will feel the effects of the eletric current on the scalp for some seconds in the begining and end of each session.
  Outcome assessors will also not be informed which group the participant is allocated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tACS+DCT (Experimental): 5 daily sessions of 30 minutes of DCT using the BrainHQ platform while simultaneously receiving theta tACS (6Hz, 1.6mA) targeting the Left Dorsolateral Prefrontal Cortex.
  Interventions: Device: Transcranial Alternating Current Stimulation; Device: Digital Cognitive Training
- SHAM+DCT (Sham Comparator): 5 daily sessions of 30 minutes of DCT using the BrainHQ platform while simultaneously receiving stimulation with the device in SHAM mode (with Ramp Up, no current during the session period and Ramp down) targeting the Left Dorsolateral Prefrontal Cortex.
  Interventions: Device: Transcranial Alternating Current Stimulation; Device: Digital Cognitive Training

INTERVENTIONS:
Device: Transcranial Alternating Current Stimulation — An alternate eletric current of 1.6mA in theta frequency is applied in the scalp, using two eletrodes (5x5cm). The eletrodes are located aiming for the left dorsolateral prefrontal Cortex area.
Device: Digital Cognitive Training — Using a tablet, the participant will do exercises that were designed to stimulate cognitive domains, especially attention and memory. In this case, we use the BrainHQ platform.

SUMMARY:
BACKGROUND Cognitive decline in older adults, especially those who develop Mild Cognitive Impairment and Alzheimer's Disease, currently has limited options of pharmacological treatments, with modest efficacy.

Digital Cognitive Training (DCT) and Transcranial Alternating Current Stimulation (tACS) are two promising tools for cognitive remediation in this population. In this exploratory study, we investigate feasibility, tolerability and preliminary effects of the association of both interventions in older adults with cognitive complaints.

METHODS Older adults with cognitive complaints are being enrolled for this study, which comprises 5 daily sessions of 30 minutes of DCT using the BrainHQ platform while simultaneously receiving theta tACS (6Hz, 1.6mA) targeting the Left Dorsolateral Prefrontal Cortex.

DETAILED DESCRIPTION:
Our goals in this study are:

* To investigate the feasibility and safety of transcranial direct current stimulation (tDCS) adjunctive to cognitive training (CT) in a cohort of individuals diagnosed with mild cognitive impairment (MCI), Subjective Cognitive Decline or Alzheimer's desease in it's initial phase (CDR 1).
* To assess the efficacy of this combined intervention in modulating cognitive function, as measured by a comprehensive neuropsychological battery.
* To explore the underlying neural mechanisms of this intervention by examining changes in event-related potentials (ERPs), specifically the N200 and P300 components, which are sensitive to cognitive processes and neural plasticity.
* To identify potential peripheral biomarkers in serum that may correlate with cognitive decline and response to the intervention.
* To determine whether the combined intervention can induce lasting changes in neurophysiological markers, as assessed by repeated ERP measurements.
* To examine the relationship between the observed cognitive improvements, alterations in neurophysiological measures, and changes in serum biomarker levels, with the aim of elucidating the biological mechanisms underlying the intervention's effects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects over 50 years old, with cognitive complaints

Exclusion Criteria:

* Estimated Intelligence Quotient <80
* Dependence on psychoactive substances (DSM-V)
* Severe psychiatric or neurological disorders
* Uncorrected visual/hearing problems
* History of syncope for an unexplained reason or seizure less than a year ago
* Previous stroke
* Use of anticoagulants
* Intracranial metallic prosthesis or cardiac pacemaker
* Any contraindication to performing tACS

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
MONTREAL COGNITIVE ASSESSMENT (MOCA) | 1 week after intervention
  The MoCA, or Montreal Cognitive Assessment, is a screening tool designed to evaluate global cognitive function, covering domains such as memory, executive function, language, visuospatial abilities, and attention. Scores range from 0 to 30, with higher scores indicating better cognitive performance and a score below 26 often considered indicative of cognitive impairment.

SECONDARY OUTCOMES:
Five digits test (FDT) | 1 week after intervention
  The FDT assesses attention, processing speed, and executive function. Participants perform tasks involving numerical stimuli under timed conditions. Performance is evaluated based on accuracy and reaction time, with faster and more accurate responses reflecting better cognitive function.
Rey-Osterrieth complex figure (ROCF) | 1 week after intervention
  The ROCF evaluates visuospatial constructional abilities, visual memory, and organizational skills. Participants copy a complex figure (copy task) and later reproduce it from memory (recall task). Scores range from 0 to 36, with higher scores representing better performance and lower scores indicating impaired abilities.
Semantic and phonemic verbal fluency | 1 week after intervention
  These tasks measure verbal fluency and executive function by asking participants to generate as many words as possible within a category (semantic fluency) or starting with a specific letter (phonemic fluency) within a limited time. Higher scores indicate better fluency and cognitive flexibility, while lower scores suggest deficits in these areas.
The Rey Auditory Verbal Learning Test (RAVLT) | 1 week after intervention
  The RAVLT assesses verbal memory, including immediate recall, learning, and delayed recall, as well as susceptibility to interference. Scores vary based on the number of correctly recalled items across trials, with higher scores indicating better memory performance and lower scores reflecting poorer memory function.
Visual P300 (Event-Related Potential) | 1 week after intervention
  The P300 is an electrophysiological measure of cognitive processing, typically recorded using EEG during an oddball paradigm. It reflects attention and working memory processes, with shorter latencies and higher amplitudes indicating more efficient neural processing and longer latencies or reduced amplitudes suggesting impairment.
Serum GFAP Analysis | before intervention
  Glial fibrillary acidic protein (GFAP) is a biomarker of astrocytic activation and neuroinflammation. Higher serum GFAP levels may indicate glial activation or neurodegeneration, while lower levels are associated with normal brain health.
Serum Beta-Amyloid Analysis | before intervention
  This analysis quantifies beta-amyloid peptides, key biomarkers of Alzheimer's disease pathology. Elevated beta-amyloid levels or an altered ratio of amyloid-beta 42/40 in serum may reflect early neurodegenerative processes, while normal levels are indicative of typical brain function.
Serum Tau Protein Analysis | before intervention
  Serum tau protein levels reflect axonal injury or neurodegeneration. Elevated tau concentrations may indicate pathological processes such as Alzheimer's disease or other neurodegenerative disorders, while normal levels suggest no significant axonal damage.
Prosaccade Task (Eye Tracking) | 1 week after intervention
  This task evaluates basic saccadic eye movement control. Participants are instructed to fixate on a peripheral target as it appears. Key metrics include reaction time, accuracy, and velocity of saccades, with faster and more accurate responses indicating better ocular motor control.
Antisaccade Task (Eye Tracking) | 1 week after intervention
  This task assesses inhibitory control and executive function. Participants must suppress a reflexive saccade to a peripheral target and instead look in the opposite direction. Metrics such as error rates, reaction times, and corrected errors are analyzed, with fewer errors and faster reaction times indicating better inhibitory control and executive function.
Visual Search Task (Eye Tracking): | 1 week after intervention
  This task evaluates visual attention and search efficiency. Participants identify a target among distractors under varying levels of complexity. Performance is measured by reaction time and accuracy, with faster and more precise responses indicating better attentional control and visual search ability.

CONTACTS AND LOCATIONS:
Overall Officials: Rogerio Panizzutti, Professor, Principal Investigator — UFRJ
Locations (1):
- Clínica da Memória - IPUB / UFRJ, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Yes
All study outcomes, including primary and secondary endpoints, will be made available upon request.
Time Frame: De-identified individual participant data (IPD) collected during the study will be made available upon reasonable request. Researchers interested in accessing the data may contact the principal investigator by providing a detailed proposal outlining the purpose of the request and intended analyses. Access will be made available upon request for a period of 5 years following the publication of the study's primary results.
Access Criteria: Data will only be shared for research purposes that align with ethical guidelines and after appropriate data-sharing agreements are established.